CLINICAL TRIAL: NCT02505126
Title: A Randomized Double-blind Clinical Trial on the Efficacy of Transcranial Direct Current Stimulation (tDCS) in Reducing Alcohol Consumption in Non-abstinent Patients With Alcohol Use Disorder
Brief Title: A Clinical Trial on the Efficacy of tDCS) in Reducing Alcohol Consumption in Non-abstinent Patients (REDSTIM)
Acronym: REDSTIM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TROJAK PHRC N 2014
Record Dates: First submitted 2015-07-15; First posted 2015-07-22 (Estimated); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Alcoholic Intoxication, Chronic
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active tDCS group (Experimental): Active tDCS
  Interventions: Device: Active tDCS
- Placebo tDCS group (Placebo Comparator): Placebo tDCS : Inactive tDCS
  Interventions: Device: Placebo tDCS

INTERVENTIONS:
Device: Active tDCS — One daily session (13:20:13) : active current flows continuously twice for 13 minutes with a rest interval (no stimulation) of 20 min 5 sessions (once a week for 5 consecutive days)
  Arms: Active tDCS group
Device: Placebo tDCS — One daily session (13:20:13) : inactive current flows continuously twice for 13 with a rest interval (no stimulation) of 20 min 5 sessions (once a week for 5 consecutive days)
  Arms: Placebo tDCS group

SUMMARY:
The study evaluates the efficacy of 1 week of tDCS (5 sessions) placebo in reducing alcohol consumption within the 24 weeks following the treatment in non-abstinent patients with alcohol use disorders versus placebo.

DETAILED DESCRIPTION:
340 patients are expected and randomized in two groups: 170 patients with active tDCS and 170 patients with placebo tDCS

Visit 1 : Patients will received one daily session (13:20:13) during 5 consecutive days: current flows continuously twice for 13min with a rest interval (no stimulation) of 20 min.

Visit 1 to 7 : Change from baseline to week 24 in Total Alcohol Consumption (TAC) and Number of Heavy Drinking Days (HDD) will be evaluated in each group.

Evaluation on alcohol consumption (daily drinking diary, alcohol craving and severity) and other assessments like mood, quality of life, safety.

The co-primary outcome of change from baseline in total alcohol consumption AND reduction in number of heavy drinking days at 6 months after treatment and its association with tDCS will be analyzed under the intention-to-treat principle using a mixed model repeated measures (8 times).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have signed and dated the informed consent form
* Male and female patients over 18 years of age
* Patients who meet at least two criteria for Alcohol Use Disorder as defined in the Diagnostic and statistical Manual of mental disorder (DSM-5)
* Patients who are motivated to reduce their alcohol consumption
* At least one attempt to achieve abstinence (unsuccessful or relapse) or to reduce alcohol consumption

Exclusion Criteria:

* Breath-alcohol concentration > 0 milligrams per litre of exhaled air at randomization (visit 1)
* < 6 heavy drinking days in the 4 weeks before randomization (European Medicines Agency, 2010; a day with alcohol consumption ≥ 60 g for men and ≥40 g for women)
* An average alcohol consumption below medium risk level according to World health Organization (WHO) in the 4 weeks before screening (WHO, 2000; ≤40g/day for men; ≤20g/day for women),
* More than 3-days abstinence prior to screening and randomization (screening visit and visit 1)
* A Revised Clinical Institute Withdrawal Assessment for Alcohol score ≥ 10 (indicating the need for medication supported detoxification) at randomization (visit 1)
* Concomitant treatment with disulfiram, acamprosate, topiramate, baclofen, naltrexone, and nalmefene (<1 month)
* History of pre-delirium tremens and delirium tremens
* DSM-5 substance use disorder other than alcohol or nicotine use disorder
* Acute psychiatric disorders that have required hospitalisation and/or immediate adjustment of psychotropic medications
* Major depression, as defined by Hamilton Depression (HDRS) scale greater than or equal to 24
* Recent change in psychotropic medication (< 1 month)
* Severe chronic psychiatric disorders including schizophrenia, paranoia and bipolar disorder type I and II
* Advanced liver, kidney, cardiac, or pulmonary disease or other acute serious or unstable medical condition that would compromise patient's participation in the study according to physician's judgment
* Contra-indications to tDCS: metal in the head, implanted brain medical devices
* Women who are pregnant or lactating
* Women of childbearing potential with a positive urine β-human chorionic gonadotrophin pregnancy test at randomization (visit 1)
* Concurrent participation in other trial
* Employees of the investigator or trial site
* Patients protected by law
* Persons who are not covered by national health insurance
* Patients, in the opinion of the investigation, not able to complete the TLFB and to complete their daily alcohol consumption in a diary (derived from the TLFB) during the 3 months of the study.
* Patients who refused to sign "safety" agreement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 339 (Actual)
Dates: Start 2015-11-23 (Actual); Primary Completion 2021-12-23 (Actual); Study Completion 2021-12-23 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 24 in Total Alcohol Consumption (TAC) | 24 weeks following the treatment
  Baseline was defined as alcohol consumption during the 28 days before randomization (visit 1). Baseline will be determined using TLFB (alcohol Timeline Follow-Back), a validated method that retrospectively obtains estimates of daily drinking using a calendar.
  TAC was defined as mean daily alcohol consumption over 28 days (in g/day)
Change from baseline to week 24 in Number of Heavy Drinking Days (HDD). | 24 weeks following the treatment
  HDD was defined as more than 60 grams of pure alcohol in men and 40 grams in women

SECONDARY OUTCOMES:
Proportion of subjects with a significant categorical shift in World health organization (WHO) risk levels of drinking | Change from baseline during the entire treatment period, and then for each 4-week period after the treatment up to week 24
  low risk (Men≤40g/d ; Women≤20g/d), medium risk (Men≤60g/d; Women≤40g/d), high risk (Men≤100g/d; Women≤60g/d, very high risk (Men>100g/d; Women>60g/d; WHO, 2010)
Proportion of subjects with a 50%, 70% and 90% reduction in alcohol consumption as well as the proportion of patients achieving maintained abstinence (cumulative abstinence duration) | Change from baseline during the entire treatment period, and then for each 4-week period after the treatment up to week 24
Change in the level of alcohol dependence severity | Change from baseline during the entire treatment period, and then for each 4-week period after the treatment up to week 24
  measured by the Alcohol Dependence Scale (ADS)
Change in craving/urge to drink assessment | Change from baseline during the entire treatment period, and then for each 4-week period after the treatment up to week 24
  using Visual Analogue Scale (VAS) the Obsessive Compulsive Drinking Scale (OCDS)
Change in Clinical Global Impression-Severity (CGI-S) and Improvement (CGI-I) | Change from baseline during the entire treatment period, and then for each 4-week period after the treatment up to week 24
Number of patients with Adverse Events (AEs) | during the entire treatment period, and then for each 4-week period after the treatment up to week 24
Change in Quality of Life | Change from baseline at week 4, week 12, and week 24 after the treatment
  SF 12
Change in validated biochemical alcohol consumption markers | Change from baseline at week 4, week 12, and week 24 after the treatment
  Gamma Glutamyl transferase (GGT), Mean Corpuscular Volume (MCV), Aspartate Aminotransferase (ASAT), Alanine Aminotransferase (ALAT) and Carbohydrate Deficient Transferrin (CDT%)
Change in scores for anxiety and depression scales | Change from baseline at week 4, week 12, and week 24 after the treatment
  Hamilton Depression Rating Scale (HDRS-21)
For smokers: change in number of cigarettes smoked/day and craving for tobacco | Change from baseline at week 4, week 12, and week 24 after the treatment
  Visual Analogue Scale (VAS), Tobacco Craving Questionnaire (TCQ),
Change in cognitive assessment | Change from baseline at week 4, week 12, and week 24 after the treatment
  Montreal Cognitive Assessment (MOCA)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France

REFERENCES:
- [Derived] Trojak B, Soudry-Faure A, Abello N, Carpentier M, Jonval L, Allard C, Sabsevari F, Blaise E, Ponavoy E, Bonin B, Meille V, Chauvet-Gelinier JC. Efficacy of transcranial direct current stimulation (tDCS) in reducing consumption in patients with alcohol use disorders: study protocol for a randomized controlled trial. Trials. 2016 May 17;17(1):250. doi: 10.1186/s13063-016-1363-8. PMID 27188795